CLINICAL TRIAL: NCT06630364
Title: A Randomized Clinical Trial Comparing Ketamine and Fentanyl for Postoperative Pain Management and Emergence Delirium Following Pediatric Tonsillectomy and Adenoidectomy
Brief Title: Comparing Ketamine and Fentanyl in Pediatric Tonsillectomy: Pain Control and Emergence Delirium Outcomes (KVFPT)
Acronym: KVFPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Yunus Oktay Atalay, MD, Prof, DESAIC, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-4354Karar651; Istanbul Medipol University (Registry Identifier: Istanbul Medipol University)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Pain, Acute; Emergence Delirium
Keywords: Tonsillectomy, Adenoidectomy, Postoperative pain management, Emergence delirium, Ketamine, Fentanyl
MeSH Terms: conditions — Pain, Postoperative; Emergence Delirium | interventions — Ketamine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Ketamine group) (Active Comparator): The patients in this group will have intravenous ketamine (0.5 mg/kg) during induction
  Interventions: Drug: ketamine
- Group II (Fentanyl Group) (Experimental): The patients in this group will have intravenous fentanyl (1 µg/kg) during induction
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: ketamine — Induction: Sevoflurane in N2O/O2, Propofol (1-1.5 mg/kg) Analgesia: Ketamine (0.5 mg/kg) Maintenance: Sevoflurane
  Arms: Group I (Ketamine group)
Drug: fentanyl — Induction: Sevoflurane in N2O/O2 Analgesia: Propofol (1-1.5 mg/kg), Fentanyl (1 µg/kg) Maintenance: Sevoflurane
  Arms: Group II (Fentanyl Group)

SUMMARY:
This study is designed to compare the effectiveness of two medications, ketamine and fentanyl, in managing pain and preventing delirium in children aged 3 to 8 years who are undergoing tonsillectomy and adenoidectomy surgery. The study aims to determine which medication is better at reducing pain and preventing delirium after surgery, and which one results in faster recovery times and fewer side effects. Children participating in the study will be randomly assigned to receive either ketamine or fentanyl during their surgery. The study will measure pain levels, recovery times, and any side effects experienced by the children. The results of this study will help doctors and anesthesiologists make better decisions about which medication to use for pain management in children undergoing tonsillectomy and adenoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 8 years
* Scheduled for tonsillectomy and adenoidectomy
* American Society of Anesthesiologists (ASA) Physical Status I-III

Exclusion Criteria:

* American Society of Anesthesiologists' Physical Status ≥4
* Known hypersensitivity or allergy to any of the study medications (acetaminophen, ketamine, fentanyl)
* Receiving chronic opioid analgesic therapy prior to surgery
* Renal disease
* Hepatic disease
* Obesity (body mass index greater than 99th percentile for age)

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Scores | From the enrollment to 8 hours post-surgery
  Face, Legs, Activity, Cry, Consolability (FLACC) Scale Range: 0 to 10 Higher scores indicate worse pain 0 = no pain, 10 = worst possible pain (Assessment of Behavioural Score: ; 0 = Relaxed and comfortable ; 1-3 = Mild discomfort ; 4-6 = Moderate pain ; 7-10 = Severe discomfort/pain.)

SECONDARY OUTCOMES:
Incidence of Emergence Delirium Following Pediatric Tonsillectomy and Adenoidectomy | From the enrollment to 8 hours post-surgery
  Pediatric Anesthesia Emergence Delirium (PAED) Scale Range: 0 to 20 Higher scores indicate more severe emergence delirium 0 = no delirium, 20 = extreme delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol Mega University Hospital, Istanbul, Bagcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelhalim AA, Alarfaj AM. The effect of ketamine versus fentanyl on the incidence of emergence agitation after sevoflurane anesthesia in pediatric patients undergoing tonsillectomy with or without adenoidectomy. Saudi J Anaesth. 2013 Oct;7(4):392-8. doi: 10.4103/1658-354X.121047. PMID 24348289
- [Background] Michelet D, Hilly J, Skhiri A, Abdat R, Diallo T, Brasher C, Dahmani S. Opioid-Sparing Effect of Ketamine in Children: A Meta-Analysis and Trial Sequential Analysis of Published Studies. Paediatr Drugs. 2016 Dec;18(6):421-433. doi: 10.1007/s40272-016-0196-y. PMID 27688125
- [Background] Eghbal MH, Taregh S, Amin A, Sahmeddini MA. Ketamine improves postoperative pain and emergence agitation following adenotonsillectomy in children. A randomized clinical trial. Middle East J Anaesthesiol. 2013 Jun;22(2):155-60. PMID 24180163
- [Background] Alghamdi F, Roth C, Jatana KR, Elmaraghy CA, Rice J, Tobias JD, Thung AK. Opioid-Sparing Anesthetic Technique for Pediatric Patients Undergoing Adenoidectomy: A Pilot Study. J Pain Res. 2020 Nov 19;13:2997-3004. doi: 10.2147/JPR.S281275. eCollection 2020. PMID 33239908